CLINICAL TRIAL: NCT05465876
Title: A Multi-Center, Open-Label, Single-Arm Phase II Trial of Antibody Combination EVUSHELD (Tixagevimab and Cilgavimab) to Provide Passive Immunity Against COVID-19 in Vaccine Non-responsive Chronic Lymphocytic Leukemia
Brief Title: Passive Antibodies Against COVID-19 With EVUSHELD in Vaccine Non-responsive CLL
Acronym: PACE-CLL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding pulled
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3989
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Lymphocytic Leukemia; COVID-19
Keywords: EVUSHELD
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Intervention Model Description: Prospective multi-centre open-label investigator-initiated single arm descriptive phase 2 clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVUSHELD (Experimental)
  Interventions: Biological: EVUSHELD

INTERVENTIONS:
Biological: EVUSHELD — EVUSHELD is a combination of 2 monoclonal antibodies (mAbs), Tixagevimab and Cilgavimab. The single dose, is to be administered intramuscular, each mAb sequentially into the deltoid

SUMMARY:
Chronic lymphocytic leukaemia (CLL) is a common lymphoid malignancy affecting older adults. CLL patients are immunocompromised by the disease itself and by several of its therapies. It has now been shown that many CLL patients do not mount an antibody response following COVID-19 vaccination and are therefore at risk of COVID-19 infection. Furthermore, patients with hematologic malignancies are known to be at increased risk of severe infection if they do acquire COVID-19 infection.

The purpose of this trial is to document evidence of passive immunity to COVID-19 infection after EVUSHELD administration with serologic and neutralization assays at multiple post administration time points in patients with no response to standard of care vaccination to COVID-19.

This trial will include a single dose of EVUSHELD to be administered, with a 1-year follow-up period, comprising of 8 health status visits.

Blood samples will be taken at screening, baseline and at multiple health status visits over the course of the year for various antibody testing and analysis. T cell reactivity to COVID-19 epitopes will be studied at baseline and again monthly for 3 months in any participants that become infected with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of CLL according to international working group CLL criteria
2. Treatment-naïve, post treatment or on-treatment for CLL
3. Male or female ≥ 18 years of age on day of signing informed consent
4. Weight ≥ 40 kg at the screening
5. Have received at least 2 standard of care SARS-CoV-2 vaccines within the last 18 months prior to enrolment. These vaccines may include all vaccines given in Canada since the beginning of the pandemic including: Pfizer BNT162b2 (COMIRNATY®), Moderna mRNA-1273 (SPIKEVAX®), and Astra Zeneca AZD1222 (Vaxzevria®)
6. Last SARS-CoV-2 vaccination ≥28 days ago and no more than 18 months ago.
7. Participants must have a demonstrated absent or suboptimal response to standard of care SARS-CoV-2 vaccinations on screening bloodwork and will be prioritized for this study as they are deemed to be at higher risk of serious COVID-19 infection.
8. Have a performance status of 0-2 on the ECOG Performance Scale.
9. Have adequate organ function laboratory values, anytime during the screening period
10. Have a life expectancy > 6 months in the opinion of the referring hematologist.
11. Female subject of childbearing potential should have a negative serum pregnancy test prior to receiving study medication (study day 0).
12. Female participants of childbearing potential should be willing to use 2 highly effective methods of birth control or be surgically sterile, or abstain from heterosexual activity for the duration of the study (after signing consent) to prevent pregnancy. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
13. Male participants should be surgically sterile or agree to use a highly effective method of contraception for the duration of the study (after signing consent) to prevent pregnancy in their partner.
14. Participants must agree to abstain from donating blood or plasma from the time of informed consent and for one year
15. Able and willing to provide signed informed consent for the trial
16. Ability to comply with protocol requirements.

Exclusion Criteria:

1. Signs and symptoms consistent with symptomatic COVID-19 illness within 30 days of consent.
2. Prior (within 30 days), current, or planned use of any of COVID-19 convalescent plasma, other monoclonal antibodies against SARS-CoV-2 or any COVID-19 treatment, or if clinically indicated as standard of care for a COVID-19 infection, should not be administered within 14 days of the EVUSHELD administration
3. Current infection requiring treatment with antibiotics or antifungals (not including prophylactic medications given with current therapy). Note: Participants completing a course of antibiotics for acute infection 7 days prior to SD0 and who do not experience a recurrence of symptoms or fever are eligible.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Has known psychiatric or substance abuse disorders that would interfere with adherence with the requirements of the trial.
6. Previous hypersensitivity reaction following administration of a monoclonal antibody
7. Currently pregnant, lactating or breast feeding
8. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 21 days of treatment (SD0).
9. Receive a COVID-19 booster shot within 90 days of EVUSHELD administration
10. Known history of allergy to any component of the study drug formulation or its excipients
11. History of clinically significant bleeding disorder, or prior history of significant bleeding or bruising following IV infusions or venipuncture.
12. Any other significant disease, disorder, or finding that may; significantly increase the risk to the participant because of participation in the study; affect the ability of the subject to participate in the study; or impair interpretation of the study data.
13. Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Passive Immunity | 12 months
  The primary study objective is to confer passive immunity to CLL patients, so the primary outcome measurement is the proportion of of participants after EVUSHELD administration with anti-spike antibodies above the minimal level set as a standard for convalescent serum or 210 u/ml using the Roche assay

SECONDARY OUTCOMES:
Surrogate Viral Neutralization Assay | 12 months
  Serum neutralization using a surrogate viral neutralization assay levels (representing levels of EVUSHELD) at months 1-6, 9 and 12 to document longevity of protection following one-time administration of the product.
Pseudo- Viral Naturalization Assay | 12 months
  Serum neutralization with a pseudo-typed viral-like particle (pseudo-virus) neutralization assay will be completed using samples obtained from 50% of participants (i.e. 25) within each treatment group at baseline and five post treatment time points. These results will be modeled over the course of the study.
Pharmacokinetic Assessments | 12 months
  Serum pharmacokinetic levels of antibodies to the COVID-19 RBD epitope at the baseline visit and visits 1, 3, 5, 7, and 8 to provide additional supportive data documenting longevity of protection following one-time administration of the product (in a subset of patients)
COVID-19 Infection (antibodies) | 12 months
  COVID-19 infection as documented by evidence of antibodies to the nucleocapsid (NC) protein
COVID-19 Infection (RAT/PCR) | 12 months
  COVID-19 infection documented by PCR or RAT.
Symptomatic COVID-19 infection | 12 months
  Symptomatic COVID-19 infection and outcomes as documented by participant clinical symptomatology and status (hospital admission, ICU admission, or death) at conclusion of the trial
Safety of EVUSHELD | 12 months
  Safety will be evaluated at each clinical visit and will include the documentation of; any changes in grade/seriousness or severity of baseline medical history, body temperature, blood pressure, oxygen saturation, heart rate, pulse, and review of symptoms, toxicities at monthly time points. Toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE, v5.0).
Baseline T cell responses to COVID-19 as a potential predictor of breakthrough COVID-19 infections | 12 months
  T cell responses at baseline will be evaluated by COVID-19-specific LEGEND-plex cytokine detection with stratification according to participant treatment group to help understand mechanisms of viral escape in participants who do become infected with COVID after EVUSHELD administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Cente, Toronto, Ontario, Canada